CLINICAL TRIAL: NCT03409991
Title: Testing the Efficacy of Opening Doors: A Career Guidance Intervention for Individuals With Psychiatric Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Erna Sally Rogers, Principal Investigator, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3727
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Psychiatric Disorder
Keywords: Psychiatric Rehabilitation; Career Counseling
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Receives the 12-week Opening Doors group sessions, and up to 8 individual career counseling sessions.
  Interventions: Behavioral: Opening Doors
- Waitlist Control (No Intervention): Offered non-vocational classes at the Boston University Center for Psychiatric Rehabilitation, and offered the chance to attend the Opening Doors program at the end of their enrolled 12-month study period.

INTERVENTIONS:
Behavioral: Opening Doors — This project is designed as a three-stage mixed methods study to test the efficacy of a career guidance intervention for individuals with psychiatric disabilities. We are using both a randomized clinical trial design coupled with a small qualitative sub-study.
  Arms: Experimental

SUMMARY:
This project is designed to develop and test a career guidance intervention called Opening Doors (OD) expected to assist individuals with psychiatric disabilities acquire knowledge, skills, and attitudes needed to pursue and advance in their careers. This project is a three-stage mixed methods study to 1) refine and pilot-test the Opening Doors career guidance intervention, 2) conduct a randomized control trial (RCT) to test the efficacy of the intervention with a waitlist control group, and 3) conduct a qualitative and process sub-study of the critical ingredients of the OD intervention from the perspective of participants. This study takes place at the Boston University Center for Psychiatric Rehabilitation (CPR). It is hypothesized that when compared to control group participants, individuals receiving Opening Doors will report 1) higher levels of vocational and pre-vocational activities, 2) greater career adaptability, fewer dysfunctional and more functional career thoughts, 3) greater work hope when compared to the waitlist control group participants, 4) greater vocational goal attainment, and 5) improved symptoms and functioning.

DETAILED DESCRIPTION:
This project is designed as a three-stage mixed methods study to test the efficacy of a career guidance intervention called Opening Doors to improve the employability and employment trajectory of individuals with psychiatric disabilities.

Stage 1 involved a pilot-test of the Opening Doors (OD) career guidance intervention to conduct a feasibility test. In Stage 2 the investigators are conducting a randomized control trial (RCT) to test the efficacy of the intervention. Stage 3, which is a qualitative and process sub-study to understand the value of the OD intervention from the perspective of participants, is being conducted simultaneously with Stage 2 The Opening Doors Intervention: The Opening Doors intervention is a new career guidance intervention for individuals with psychiatric disabilities that uses traditional career guidance resources, progressive employment principles and mainstream Internet-based resources, delivered in the context of providing tailored supports for participants' with mental illness. Opening Doors is designed as an approximately 12- week group and individual career guidance intervention. The curriculum is delivered by trained career counselors in small groups over about 20 sessions of 90 minutes each with the addition of up to 8 weekly 1 hour individual sessions. Opening Doors also has optional on-going drop-in hours available for participants of the program (current and past) to improve their job application potential on an on-going basis. Opening Doors includes considerable peer involvement i.e. the consultation and inclusion of individuals with lived experience of psychiatric disabilities in the development and delivery of the intervention.

Method: The Opening Doors intervention has been pilot-tested using a simple pretest-posttest design in order to assess feasibility of the intervention and research procedures. The investigators are currently using a randomized clinical trial design (RCT) to test the effectiveness of the Opening Doors intervention. Up to 108 participants are expected to participate in the intervention. Baseline assessments are completed and random assignment to experimental or control conditions are performed, stratifying for gender and minority status using a computer generated randomization plan. Assessments are conducted at baseline, 3, 6, 9 and 12 months post-baseline for both experimental and control groups. Control participants are placed on a waitlist and offered participation at a later date i.e. 12 months after the baseline assessment. The investigators use qualitative methods for a sub-study and process evaluation. Twelve participants (2 per wave) who have completed at least 12 sessions of the OD will be invited to participate in one-hour qualitative interviews to obtain their perspectives on the intervention. Each participant participates in a one hour single-session audio-taped interview by research staff. Data from the qualitative interviews is collected using an interview guide and participants are probed for perceived benefits of the intervention and hypothesized helpful mechanisms of OD. The investigators also query the staff about their perceptions of the barriers and facilitators to delivering OD. Additional process information described above in "process data" is collected on all study participants.

Data Analysis: Depending on the level of measurement, analysis of variance, t-tests, or chi-square tests were conducted to determine baseline equivalency between Experimental and Control groups. All hypotheses were tested using mixed modeling analyses, adjusting for baseline values and examining effects for time, group, and the group-by-time interactions. We found no differences between the experimental and control groups using an ITT approach or adjusting for intervention intensity. We conducted responder analyses to further explore what worked and for whom.

ELIGIBILITY:
Inclusion Criteria:

1. are 18 years or older;
2. have a psychiatric disability as evidenced by a) the presence of a psychiatric diagnosis, b) the interference of psychiatric symptoms with important areas of life functioning such as, work or school, and c) current or past use of psychiatric services such as, medications, hospitalizations, psychotherapy, etc.;
3. express an interest in exploring their career options;
4. are unemployed or engaged in part-time employment;
5. express an interest in working in the future;
6. have basic knowledge of using computers; and,
7. are willing and able to attend a 1-2 hour orientation session at the Recovery Center.

Exclusion Criteria:

1. are unable to give full and knowing consent;
2. are unable to participate in data collection;
3. are actively receiving vocational counseling; and, 4) have full-time paid employment;

5) have a legal guardian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2015-09-24 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Employment and Vocational Activities Checklist | 12 months
  Participants will report greater engagement in vocational activities. Employment and Vocational Activities Checklist, a brief instrument used in prior Center studies that inquires about current pre-employment and vocational activities, including for example, career development activities and independent job searches
Work Hope Scale (Juntunen & Wettersten, 2006) | 12 months
  24-item 7-point Likert-type scale that measures the construct of work hope, and includes: Work Goals, Agency, and Pathways. The scale is a stable and well-validated measure with reported internal consistency of the overall scale of .93 and .87, .68 and .81 for the sub-scales
Goal Attainment Scale (GAS, Kiresuk, et al, 1968) | 12 months
  Goal Attainment Scale provides a structured approach to determining goal achievement regardless of the type or uniqueness of goal (Kiresuk & Sherman, 1968). Recent reviews of GAS confirms that it can be useful in measuring rehabilitation goals, is reliable and sensitive to change (Marson, et al., 2009; Hurn, et al., 2006, Turner-Stokes, 2009)
Career Adapt-Abilities Scale (CAAS; Savickas & Porfeli, 2012) | 12 months
  Career Adapt-Abilities Scale (CAAS; Savickas & Porfeli, 2012) measures an individual's psychosocial readiness and resources for coping with current and imminent vocational development tasks, occupational transitions, and work traumas using four scales which measure concern, control, curiosity, and confidence. Internal consistency estimates for the subscale and total scores ranged from good to excellent i.e. .82 to .88. Concurrent validity evidence was found to be strong between the subscales of CAAS and the Vocational Identity Status Assessment (VISA; Porfeli, Lee, Vondracek, & Weigold, 2011)
Career Thoughts Inventory (CTI; Sampson et al., 1996) | 12 months
  The CTI consists of 48 Likert-scale items rated on a 4-point agree scale representing typical dysfunctional/negative career thoughts including Decision-Making Confusion, Commitment Anxiety, and External Conflict. The CTI developers report alpha coefficients for the total score ranging from .93 to .97; and for the subscales ranged from .74 to .94. The authors also provide support for the CTI's construct validity, convergent validity, and criterion validity.
Behavior and Symptom Identification Scale (BASIS - 24) (Eisen, et al., 2004, Eisen et al., 2006) | 12 months
  The BASIS-24 is designed to measure mood disturbances, anxiety, interpersonal and role functioning, daily living skills, psychotic symptoms, impulsivity and substance use using a 5-point Likert-type scale. Extensive and excellent reliability and validity data exists for the instrument from a national study involving over 5,000 participants (Eisen, et al., 2004; Eisen, et al., 2006)
Brief Quality of Life Scale, Subjective Items (Lehman Quality of Life Scale, Brief Version, Lehman, 1988) | 12 months
  Brief Quality of Life Scale, Subjective Items (Lehman Quality of Life Scale, Brief Version, Lehman, 1988) measures both objective and subjective quality of life across multiple domains including living situation, family relations, social relations, work, and the like. It has considerable psychometric data suggesting adequate validity and reliability (Lehman, 1995; Russo et al., 1997). We will employ 2 items from this scale: the subjective measures of life in general and work satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Erna S. Rogers, Sc.D., Principal Investigator — Boston University Center for Psychiatric Rehabilitation
Locations (1):
- Boston University Center for Psychiatric Rehabilitation, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT03409991/ICF_000.pdf